CLINICAL TRIAL: NCT02179983
Title: A Randomized Controlled Trial of Pulmonary Rehabilitation After Exacerbations of Bronchiectasis
Brief Title: Tayside Rehabilitation in Bronchiectasis Exacerbations (TRIBE) : a Randomized Controlled Trial
Acronym: TRIBE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHSTayside
Record Dates: First submitted 2014-06-29; First posted 2014-07-02 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; rehabilitation; exercise; exacerbations
MeSH Terms: conditions — Bronchiectasis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Standard care for exacerbation and follow-up without rehabilitation
- Pulmonary rehabilitation (Experimental): 6 weeks of exercise and patient education after exacerbation (pulmonary rehabilitation)
  Interventions: Procedure: Pulmonary rehabilitation

INTERVENTIONS:
Procedure: Pulmonary rehabilitation — 6 weeks of supervised exercise and education (pulmonary rehabilitation)
  Arms: Pulmonary rehabilitation
Procedure: Pulmonary rehabilitation — 6 weeks of exercise and patient education following exacerbation (pulmonary rehabilitation)
  Arms: Pulmonary rehabilitation

SUMMARY:
Pulmonary rehabilitation is well established as a treatment in COPD. After exacerbations of COPD, rehabilitation is associated with reduced frequency of exacerbations and improved exercise capacity. No data are available in bronchiectasis.

This study will randomly assign patients with bronchiectasis exacerbations to pulmonary rehabilitation or standard care. The hypothesis is that exercise capacity will be improved by pulmonary rehabilitation at 8 weeks.

DETAILED DESCRIPTION:
Background: Pulmonary rehabilitation is an effective treatment after exacerbations of COPD to prevent future exacerbations and to improve breathlessness and quality of life. Its effectiveness after exacerbations of bronchiectasis has never been demonstrated.

Aims: To determine if a 6 week course of pulmonary rehabilitation improves exercise capacity at 8 weeks after exacerbation.

Study Design: Randomised controlled trial. Methods: The study will take place in NHS Tayside. 40 patients with a history of bronchiectasis confirmed by HRCT will be included. Patients will be monitored using diary cards for exacerbations. At the onset of an exacerbation patients will be treated with a standard 14 day course of antibiotic therapy and randomised to one of two arms: Pulmonary rehabilitation or standard care. Patients randomised to pulmonary rehabilitation will undergo a 6 week course of supervised pulmonary rehabilitation. Patients will undergo study assessments (6-minute walk test, Quality of life questionnaires, pulmonary function tests (FEV1, FVC, FEF 25-75), symptoms recorded by symptom diaries and sputum microbiology).Assessments will be performed at the start and end of exacerbations, at 6-8 weeks post exacerbation (after completion of pulmonary rehabilitation in patients randomised to rehabilitation) and at 12 weeks.

Outcome: The primary outcome is 6 minute walk distance at 8 week post exacerbation Expected Conclusion: We will determine the effectiveness of pulmonary rehabilitation after exacerbations of bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

Bronchiectasis confirmed on High Resolution CT scan Clinical Bronchiectasis confirmed by a respiratory physician. Documented exacerbation within the last year. Independently mobile - i.e. able to undertake pulmonary rehabilitation

Exclusion Criteria:

* Inability to give informed consent to participate
* Age <18 years
* Primary diagnosis of Chronic Obstructive Pulmonary Disease
* Significant comorbidity that would limit the ability to undertake pulmonary rehabilitation - i.e. Cerebrovascular, cardiovascular or musculoskeletal disease.
* Cystic Fibrosis
* Aortic aneurysm
* Recent myocardial infarction (within previous year)or unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance | 8 weeks post exacerbation

SECONDARY OUTCOMES:
Time to next exacerbation | 6 months
The Quality of life | 8 weeks and 12 weeks
  St Georges respiratory questionnaire COPD assessment test
Pulmonary function tests | 8 weeks and 12 weeks
  Pulmonary function tests (FEV1, FVC, FEF25-75)
Respiratory symptoms | 8 weeks and 12 weeks
  Patient diary cards
Sputum microbiology | 8 weeks and 12 weeks
  Proportion of patients with positive sputum microbiology of potential pathogenic microorganisms (Haemophilus influenzae, Pseudomonas aeruginosa, Moraxella catarrhalis, enterobacteriaceae) versus patients without sputum colonisation.
6 minute walk distance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James D Chalmers, MBChB, PhD, Principal Investigator — NHS Tayside; Tom Fardon, MD, Principal Investigator — NHS Tayside
Locations (1):
- Clinical Research Centre, University of Dundee, Dundee, United Kingdom

REFERENCES:
- [Derived] Chalmers JD, Crichton ML, Brady G, Finch S, Lonergan M, Fardon TC. Pulmonary rehabilitation after exacerbation of bronchiectasis: a pilot randomized controlled trial. BMC Pulm Med. 2019 May 6;19(1):85. doi: 10.1186/s12890-019-0856-0. PMID 31060529